CLINICAL TRIAL: NCT03880383
Title: BRIGHT Coaching: A Randomized Controlled Trial on the Effectiveness of a Developmental Coach System to Empower Families of Children With Emerging Developmental Delay
Brief Title: BRIGHT Coaching Program for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Alberta (Other)
Responsible Party: Principal Investigator, Annette Majnemer, Professor - School of Physical & Occupational Therapy. Vice Dean - Education, Faculty of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-3159
Record Dates: First submitted 2019-03-10; First posted 2019-03-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Wellness 1; Parent-Child Relations; Child Developmental Delay; Parenting; Parent-child Problem; Child Development Disorder; Autism Spectrum Disorder
Keywords: brain-based developmental disorders; child development; preschool skills and development; parenting stress; parenting mental health; coaching intervention; online education; parent peer support; developmental delay
MeSH Terms: conditions — Learning Disabilities; Developmental Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm pragmatic randomized controlled trial (RCT) comparing a developmental coaching and e-health services intervention plus usual and locally available care to the control state in which children and their families receive usual and locally available care over an 18-month time frame. The control group will be provided with partial intervention at the end of the 18 month study. The target population for this novel service delivery model is families with children aged 1.5 to 4.5 years old with developmental concerns, who are beginning to manifest impairments in developmental domains (e.g. motor, cognitive, speech, social and/or behavioural).
Masking Description: In the context of the provided intervention (coaching vs. usual and locally available care) and outcome measures used (self-reported),blinding of participants, care providers, investigators nor that of the assessor is possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Coaching (Experimental): Upon enrollment to the study, parents in this group will have immediate access to the full intervention:
  * Coaching: Telephone contact with coaches, who will provide information, education and support about the child's development. Coaching will be adapted to family needs, situation, preferences and child's condition.
  * Online parent education: Parents will be provided access to empowering online tools, such as educational resources, chosen or developed by other parents and researchers.
  * Peer support tools: Parents will have access to a secure online social media tool to connect to other parents going through a similar experience. Through this tool, parents can help support each other, and share their experiences and knowledge.
  Interventions: Behavioral: Coaching; Behavioral: Online parent education; Behavioral: Online peer support
- Group 2- Partial and delayed coaching (Other): Parents in this group will have delayed and partial access to coaching, at the end of the 18-month period. Parents in this group will have a one-time session with a developmental coach who can give them guidance about their child's development. Parents in this group will also then get access to online parent education and peer support tools, indefinitely, until the online platform is de-activated.
  * Both arms/groups* will obtain usual care for their child, in addition and independent of full or partial coaching.
  Interventions: Behavioral: Online parent education; Behavioral: Online peer support

INTERVENTIONS:
Behavioral: Coaching — Parents will interact and communicate regularly with a coach in person or by telephone. Coaches will be responsible for: identifying developmental concerns, proactive health promotion, guidance and training for developmental stimulation, parent support and education about child development, navigation of the health care system and self-management techniques. The frequency of coaching will be: once a month (minimum), for 18 months, at an average of 2.5 hours per month.
  Other Names: coaching, family support
  Arms: Group 1 - Coaching
Behavioral: Online parent education — Parents will be provided access to an online platform which will provide educational resources and access to parent-parent support. Online resources on child development are curated by researchers and representative of parent groups, and linked to this online platform. The themes covered in the online tool include resources on child development, accessing health care services and managing emotions and family dynamics. These topics range from: practical tips for managing day-to-day challenges, strategies to cope and support the child's transitions from one stage to another, practical tips when looking for developmental services for the child: knowing where and how to access services.
  Other Names: educational resources
Behavioral: Online peer support — Parents will have access to a secure online social media tool to connect to other parents going through a similar experience. Through this tool, parents can help support each other, and share their experiences and knowledge. This will put each family at the centre of each network (family, friends, health providers), allowing family networks to link with one another. Families will be able to find resources, create connections with the coach, health providers and other families, thus creating a network to support one another.
  Other Names: parent support, patient support, sharing experiences

SUMMARY:
Children with, or at elevated risk for, brain-based developmental disabilities can experience lifelong consequences and challenges throughout their development. In particular, preschool years (3-6 years of age) can be stressful as families wait to get services and care for their child. Nationally and internationally, service delivery models during this critical period are not standardized, and differ within and across provinces and across patient conditions, leading to long wait times, service gaps and duplications.

This study has two main hypotheses:

1. A standardized approach to "coaching" (i.e. coach + online education tools + peer support network) is feasible in the real-life context, and acceptable to caregivers and can be delivered across multiple sites in urban/suburban/rural settings.
2. A standardized approach to "coaching" enhances parental health (parents' empowerment and sense of competence, quality of life, and minimizes parenting stress), family health care experience (care coordination experience and process of care) at similar health care cost (economic analysis), when compared to usual and locally available care.

DETAILED DESCRIPTION:
Rationale:

Children with, or at elevated risk for, brain-based developmental disabilities experience chronic lifelong functional consequences with new challenges emerging at each stage of development. In the preschool years (3-6 years), needs arise from vulnerabilities linked to critical and newly emerging cognitive, speech, motor, behavioural and social skills. The preschool years are a time of stress for families as young child awaits assessment, or even as they receive services for brain-based disorders. Similarly, the system and society struggle to meet needs of families in a timely and appropriate manner in the face of escalating costs. Given these struggles, there is a need to examine whether a health-coach style of intervention coupled with parent education delivered through an online platform can be effective in empowering families, by delivering information, providing social (parent to parent) supports, and decreasing demand on health and developmental services. This innovation provides a significant service re-design in a system at critical point of transition.

Study objective:

To evaluate the feasibility and the effectiveness (changes in parent health, developmental service utilization and cost effectiveness) of a self-management intervention (including developmental coach, online education tools and support network), when compared to usual and locally available care in service delivery practices, for parents of preschool children with suspected developmental delays.

Methodology / Study design:

This is a prospective, two-arm pragmatic randomized controlled trial (RCT) comparing a developmental coaching and e-health services intervention plus usual care to the control state in which children and their families receive usual and locally available care over an 18-month time frame. The target population for this novel service delivery model is children aged 1.5 to 4.5 years old who are at a high risk for or suspected of having developmental delays, that are beginning to manifest impairments in developmental domains (e.g. motor, cognitive, speech, social and/or behavioural). In the first year, a technology-supported health coach service delivery model will be developed in conjunction with families. A feasibility/acceptability pilot study was conducted to ensure that the intervention is feasible in the real life context across 4 participating Canadian provinces.

Participants:

Eligible children and their families will be recruited to include children who are 1.5 to 4.5 years at the age at enrolment. Children will be living in four diverse parts of Canada to ensure national representation and future scalability: Vancouver; Winnipeg; Montreal and Halifax. Participants' postal codes will be analyzed to ensure representation: rural/remote, small urban and large urban/metro representation with purposeful sampling as required. From the patient population perspective, two different groups that are likely to manifest new global developmental delays at this stage will be recruited. They are at high risk for brain-based developmental delays, however some will have no delay and others will have mild, moderate or severe delays.

Study procedures: Intervention and control Recruitment begins with family contact. Families are contacted via the centre to which they were referred for developmental diagnosis and assessment. A member of the clinical team will ask if they are interested to learn more about the BRIGHT Coaching study. If interested, the families' contact information will be shared with the local research assistant (RA) overseeing the trial. The RA will speak to a parent by phone and follow up with an introductory letter by mail explaining the procedures of the study, together with the consent form and a self-addressed stamped envelope to return to the RA if interested in participating. After 2 weeks, if no consent form is received, the RA will call the family once again to determine their interest in participating. Once consent is signed, participants will conduct baseline assessments including documentation of their care and social networks, and be randomized using a computer-generated algorithm; randomization will be stratified by site. The allocation ratio for intervention or control will be 1:1 for each site.

ELIGIBILITY:
Children are beginning to manifest delays in one or more domains of development, and they have been newly referred to a service to get assessed, diagnosed, and/ or for therapeutic intervention. Their families are thus in the early stages of their journey of getting assessment, diagnosis and/or intervention.

Inclusion Criteria:

* Children between the ages of 1.5 years to 4.5 years at enrolment;
* Suspected or confirmed delays in one or more developmental domains (such as motor, cognitive, speech, social and/or behavioural).
* Has been newly referred to a given service agency/program for assessment and/or intervention services (some services may have been provided in the past in infancy)
* Willing to participate in the study for 3 assessments: at enrolment; 8 months later, and 12 months later.

Exclusion Criteria:

* Non-English or non-French speaking;
* Unwilling or unable to participate in intermittent assessments (by phone or in-person).
* Do not have access on a routine basis to the internet through a desktop, laptop or mobile.

Ages: 18 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Family Empowerment Scale (FES) - change is being assessed. | 10-15 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  The FES is composed of 34 statements that describe how a parent or caregiver of a child with an emotional, behavioral and/or developmental challenges may feel about his or her situation (i.e. sense of empowerment). For each statement, the participant is asked to circle the response that best describes how the statement applies to him/her. The scale ranges from 1 (Not True at All) to 5 (Very True), for a maximum of 170 points and a minimum of 34 points. A higher score represent a higher sense of empowerment (i.e. better outcome).
Parent Sense of Competency (PSOC) Scale - change is being assessed. | 10-15 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  The PSOC measures parents' sense of competence and is a 17-item scale, with 2 subscales. Each item is rated on a 6-point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". A higher score indicates a higher parenting sense of competency.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) - change is being assessed. | 7-10 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  36-question survey about parental well-being and health-related quality of life. The following domains are being assessed: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Participant is asked to rate his/her ability for each statement as "Yes, Limited a lot", "Yes, Limited a Little", or "No, Not Limited at all". The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100; Lower scores = more disability, higher scores = less disability.
Parenting Stress Index - 36 (PSI-36) - change is being assessed. | 7-10 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  The PSI is a self-report screening tool that helps providers and families identify the sources and different types of stress that come with parenting. Parents report their level of agreement with 36 items that fall into three subscales:
  * Parental Distress (PD)-The extent to which parents feel competent, restricted, conflicted, supported, and/or depressed in their role as a parent.
  * Parent-Child Dysfunctional Interaction (P-CDI)-The extent to which parents feel satisfied with their child and their interactions with them.
  * Difficult Child (DC)-How a parent perceives their child to be, whether the child is easy or difficult to take care of.
  * Total Stress-indication of overall level of stress a person is feeling in their role as a parent.
  For most items, parents should respond by circling SA (strongly agree), A (agree), NS (not sure), D (disagree), SD (strongly disagree). Raw scores are added and higher scores represent higher stress levels.
Measure of Process of Care - 20 (MPOC - 20) - change is being assessed. | 10 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  20-item survey measuring the extent to which care is family-centred. Participants need to select one option (ranging from 0-7 or "Not applicable" to "A very great extent") that best applies to them for each statement. Raw scores are being summed (for a maximum of 140 points and a minimum of 0 points) and higher scores represent higher perceived family-centred care that the family is receiving.
Resource Utilization Questionnaire - Preschoolers (RUQ-P) - change is being assessed. | 45 minutes at each study visit (at baseline, 8 months post-entry [immediately post-intervention], 12 months post-entry [follow-up])
  The RUQ-P collected data on resource use; service intensity; and out-of-pocket costs, such as hourly rates, costs of materials, and travel costs. The following services/resources are being assessed: Speech-Language or Communication Services; Occupational Therapy; Physiotherapy; Child-focused recreational activities; Intervention/Consultation for Challenging Behaviour; Structured/Systematic Teaching with Specific Goals (Optional); Relationship-Based Intervention ; Medication/Supplements and Special diet; Visits with additional Health Professionals; Parents' Use of Health Services and Medications and Other Resources; Purchased Materials, Equipment, etc.; Respite; Time Associated with Treatment and Care; Government Tax Rebates, Deductions, Subsidies and Other Supports; Insurance Plan. For each question/statement, a multiple choice of responses are provided and participant is asked to select one. Responses are analysed using descriptive statistics (frequencies of selected answers).

OTHER OUTCOMES:
Vineland Adaptive Behavior Scales (Vineland) | 20-60 minutes, at baseline visit only.
  The Vineland is a survey that is conducted with parents or caregivers, measuring 4 domains of the child's adaptive behaviour (with 2-3 subdomains in each): the child's communication, daily living skills, socialization and motor skills. Eleven general subdomains are grouped into those four main domains. The scores of the subdomains are added to form the domain composite scores. The four domain composite scores then combine to form the adaptive behaviour composite.
  Scoring: Each subdomain question is scored on a 3-point scale: score of 2 refers to "Usually", 1 refers to "Sometimes" and 0 refers to "Never". Higher scores indicate better outcome (i.e. higher adaptive behaviour in each domain).
  The following interpretation tools/scores are provided: 1) Domains and Adaptive Behaviour Composite: Standard scores (M = 100, SD = 15), percentile ranks, adaptive levels. 2) Subdomain: V-scale score (M = 15, SD = 3), Adaptive levels, age equivalents.
Readiness to receive coaching | 5 minutes, at baseline visit only.
  This eight-question/statement screening tool was developed in-house to assess the participants' readiness to receive the coaching intervention. Each statement (e.g. "I am willing to talk, engage and share with my coach") will be rated on a 5-point Likert Scale ranging from "Strongly Disagree" to "Strongly Agree".
Demographic form | 10-15 minutes, at baseline visit only.
  Survey on sociodemographics and family structure/composition

CONTACTS AND LOCATIONS:
Overall Officials: Annette Majnemer, PhD, Principal Investigator — Research Institute of McGill University Health Centre; Maureen O'Donnell, MD, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (4):
- Canada (4):
  - Child Health BC, BC Children's Hospital, UBC, Vancouver, British Columbia
  - Specialized Services for Children and Youth (SSCY) Centre, Winnipeg, Manitoba
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - Research Institute of McGill University Health Centre, Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
At this time, plan has not been created

REFERENCES:
- [Background] Majnemer A, Limperopoulos C, Shevell MI, Rohlicek C, Rosenblatt B, Tchervenkov C. A new look at outcomes of infants with congenital heart disease. Pediatr Neurol. 2009 Mar;40(3):197-204. doi: 10.1016/j.pediatrneurol.2008.09.014. PMID 19218033
- [Background] Vohr B. Long-term outcomes of moderately preterm, late preterm, and early term infants. Clin Perinatol. 2013 Dec;40(4):739-51. doi: 10.1016/j.clp.2013.07.006. Epub 2013 Sep 20. PMID 24182959
- [Background] Mazer, B., Majnemer, A., and Shevell M., Service utilization and health promotion of children with neuro-developmental disabilities. Neurodevelopmental disabilities: Clinical and scientific foundation, 2009: p. p. 426-441.
- [Background] Grilli L, Feldman DE, Swaine B, Gosselin J, Champagne F, Pineault R. Wait times for paediatric rehabilitation. Healthc Policy. 2007 Feb;2(3):e171-87. PMID 19305712
- [Background] Miller AR, Condin CJ, McKellin WH, Shaw N, Klassen AF, Sheps S. Continuity of care for children with complex chronic health conditions: parents' perspectives. BMC Health Serv Res. 2009 Dec 21;9:242. doi: 10.1186/1472-6963-9-242. PMID 20025770
- [Background] Lorig KR, Sobel DS, Stewart AL, Brown BW Jr, Bandura A, Ritter P, Gonzalez VM, Laurent DD, Holman HR. Evidence suggesting that a chronic disease self-management program can improve health status while reducing hospitalization: a randomized trial. Med Care. 1999 Jan;37(1):5-14. doi: 10.1097/00005650-199901000-00003. PMID 10413387
- [Background] Leahey TM, Wing RR. A randomized controlled pilot study testing three types of health coaches for obesity treatment: Professional, peer, and mentor. Obesity (Silver Spring). 2013 May;21(5):928-34. doi: 10.1002/oby.20271. PMID 23784896
- [Background] Huffman MH. HEALTH COACHING: a fresh, new approach to improve quality outcomes and compliance for patients with chronic conditions. Home Healthc Nurse. 2009 Sep;27(8):490-6; quiz 496-8. doi: 10.1097/01.NHH.0000360924.64474.04. PMID 19745624
- [Background] Kiresuk, T.J., Smith A., and Cardillo J.E. , Goal attainment scaling: Applications, theory, and measurement. Psychology Press, 2014.
- [Background] Ottenbacher KJ, Msall ME, Lyon N. Measuring developmental and functional status in children with disabilities. Pediatr Phys Ther. 2000 Winter;12(4):198-9. No abstract available. PMID 17091034
- [Background] Abidin, R.R., PARENTING STRESS INDEX (4th ed.). 2012: Lutz, FL: PAR.
- [Background] Koren PE, D.N., Friesen BJ. , Measuring empowerment in families whose children have emotional disabilities: a brief questionnaire. Rehabilitation Psychology, 1992. 37(4): p. 305.
- [Background] Ohan JL, L.D., Johnston C., The Parenting Sense of Competence scale: Evidence of a stable factor structure and validity. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 2000 Oct. 32(4): p. 251.
- [Background] Ware JE, S.K., Kosinski M, Gandek B, SF-36 HEALTH SURVEY MANUAL AND INTERPRETATION GUIDE, M.T.H.I. Boston, New England Medical Center, Editor. 1993.
- [Background] Dyke P, Buttigieg P, Blackmore AM, Ghose A. Use of the measure of process of care for families (MPOC-56) and service providers (MPOC-SP) to evaluate family-centred services in a paediatric disability setting. Child Care Health Dev. 2006 Mar;32(2):167-76. doi: 10.1111/j.1365-2214.2006.00604.x. PMID 16441851
- [Background] Borgatti SP, E.M., Freeman LC, Ucinet for Windows: Software for Social Network Analysis, M.H.-A.T. Cambridge, Editor. 2002.
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681
- [Background] Katz P, Morris A, Trupin L, Yazdany J, Yelin E. Disability in valued life activities among individuals with systemic lupus erythematosus. Arthritis Rheum. 2008 Apr 15;59(4):465-73. doi: 10.1002/art.23536. PMID 18383406
- [Derived] Majnemer A, O'Donnell M, Ogourtsova T, Kasaai B, Ballantyne M, Cohen E, Collet JP, Dewan T, Elsabbagh M, Hanlon-Dearman A, Filliter JH, Lach L, McElroy T, McGrath P, McKellin W, Miller A, Patel H, Rempel G, Shevell M, Wittmeier K; Parent-Panel. BRIGHT Coaching: A Randomized Controlled Trial on the Effectiveness of a Developmental Coach System to Empower Families of Children With Emerging Developmental Delay. Front Pediatr. 2019 Aug 7;7:332. doi: 10.3389/fped.2019.00332. eCollection 2019. PMID 31440489

DOCUMENTS (1):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03880383/Prot_000.pdf